CLINICAL TRIAL: NCT04964518
Title: A Phase Ib/II Study of APG-2575 in Combination With Azacitidine in Patients With Acute Myeloid Leukemia (AML), Mixed Phenotype Acute Leukemia (MPAL), Chronic Myelomonocytic Leukemia (CMML) and Higher-Risk Myelodysplastic Syndrome (MDS
Brief Title: A Study of APG-2575 in Combination With Azacitidine in Patients With Acute Myeloid Leukemia (AML)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APG2575AU101
Record Dates: First submitted 2021-06-23; First posted 2021-07-16 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: AML, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Lisaftoclax

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APG2575 + Azacitidine (Experimental): 200 mg APG2575 dose ramp up +AZA
  Interventions: Drug: APG 2575 ramp up arm

INTERVENTIONS:
Drug: APG 2575 ramp up arm — APG2575 ramp up + Azacitidine
  Other Names: APG2575

SUMMARY:
This is a Phase Ib/II, open-label, multi-center study evaluating the safety, tolerability, efficacy and PK of APG-2575 in combination with Azacitidine in the patients with AML/MPAL or MDS/CMML. The study consists of dose escalation (Part I) and dose expansion phase (Part II)

DETAILED DESCRIPTION:
The patients with histologically confirmed relapsed or refractory (R/R) AML/MPAL/CMML or relapsed/refractory Higher-Risk MDS by WHO classification for which no available standard therapies are indicated or anticipated to result in a durable response will be enrolled.

This will be a 3+3 dose escalation to determine the DLTs and MTD/RP2D of APG-2575 (see dose escalation table) given in combination with Azacitidine

ELIGIBILITY:
Inclusion Criteria:

Patients with a diagnosis of histologically confirmed relapsed or refractory (R/R) acute myeloid leukemia (AML) or mixed phenotype acute leukemia (MPAL) or Chronic Myelomonocytic Leukemia (CMML) or relapsed/refractory Higher-Risk MDS by 2016 WHO classification for which no available standard therapies are indicated or anticipated to result in a durable response.

* MPAL will include biphenotypic leukemia, bilineal leukemia, undifferentiated leukemia, mixed lineage leukemia, leukemia of ambiguous lineage, T/myeloid leukemia, B/myeloid leukemia, or other diagnosis indicating the presence of multiple lineages within the cell population.
* Relapsed/refractory MDS will be defined as prior receipt of 4 cycles of HMA therapy with failure to attain a response, or progression of disease or relapse at any time after prior response to HMA therapy with Overall Revised International Prognostic Scoring System (IPSS-R) score > 3 (intermediate, high or very high).

Exclusion Criteria:

1. Pregnant women.
2. Uncontrolled intercurrent illness including, but not limited to active uncontrolled infection, symptomatic congestive heart failure (NYHA Class III or IV), unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Have had leukemia therapy within 14 days prior to starting investigational drug.

   However, patients with rapidly proliferative disease may receive hydroxyurea as needed until 24 hours prior to starting therapy on this protocol and during the first cycle of study.
4. Have taken strong inhibitors or inducers of CYP3A4 within 7 days prior to the first dose of APG-2575.
5. Have acute promyelocytic leukemia (French-American-British Class M3 AML or WHO classification APL with PML-RARA) or AML/MPAL with BCR-ABL1 positive.
6. Active infection requiring systemic antibiotic/antifungal medication, known clinically active hepatitis B or C, or HIV infection or active COVID-19. (Patients who have received COVID-19 vaccination will be considered as eligible for the study.)
7. Have active/ongoing graft-versus host disease (GVHD) or require continued treatment with systemic immunosuppressive agents (calcineurin inhibitors within 4 weeks prior to the first dose).
8. Myeloablative therapy with autologous or allogeneic hematopoietic stem cell rescue within 6 months of study treatment initiation.
9. Documented hypersensitivity to any of the components of the therapy program.
10. Active, uncontrolled CNS leukemia.
11. Men and women of childbearing potential who do not practice contraception. Women of childbearing potential and men must agree to use at least 1 form of barrier birth control (such as condom) prior to study entry and for the duration of study participation.
12. History of other malignancies within 2 years prior to study entry, with the exception of:

    * Adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast.
    * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin.
    * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intention requires discussion with sponsor.
13. Failure to have recovered (Grade > 1) from prior treatment (including chemotherapy, targeted therapy, immunotherapy, experimental agents, radiation, or surgery), except for alopecia.
14. Unable to swallow tablets or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
15. Significant screening electrocardiogram (ECG) abnormalities including left bundle branch block, 2nd degree atrioventricular (AV) block type II, 3rd degree block, or corrected QT interval (QTc) ≥470 msec.
16. Any other condition or circumstance that would, in the opinion of the investigator, make the patient unsuitable for participation in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
DLT | 28 days
  Dose-limiting toxicity (DLT) rate at each dose level
  DLT will be assessed within the first 28-day cycle of study treatment via CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Qian Niu, MD, Principal Investigator — Ascentage Pharma
Locations (9):
- United States (5):
  - UCLA Medical cetner Division of Hematology, Los Angeles, California
  - Novant Health, Charlotte, North Carolina
  - Novant Health, Winston-Salem, North Carolina
  - MDACC, Houston, Texas
  - Swedish Medical Center, Seattle, Washington
- Australia (4):
  - Pindara Private Hospital, Benowa, Queensland
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - The Northern Hospital, Epping, Victoria
  - Royal Perth Hospital, Perth, Western Aus

IPD SHARING:
Plan to Share IPD: Undecided